CLINICAL TRIAL: NCT00910013
Title: A Randomized Trial Comparing the Efficacy on Post-operative Analgesia of Intra-articular Ropivacaine Added to a Femoral Block After Total Knee Replacement
Brief Title: Femoral Block With or Without Ropivacaine for Analgesia After Total Knee Replacement (TKR)
Acronym: TKR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hopital de l'Enfant-Jesus (Other)
Responsible Party: Dr Stéphane Pelet, MD, PhD, Département orthopédie, CHA-Pavillon Enfant-Jésus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEJ-340
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2009-05

CONDITIONS: Total Knee Replacement
Keywords: TKR; Femoral block; Ropivacaïne; intra-articular ropivacaïne; post-operative analgesia
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ropivacaine + femoral block (Experimental): After the surgery is proceeded and after the closure of the joint capsule, 20 cc of ropivacaine 0.5% is inserted intra-articular through a catheter.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — 0.5% intra-articular ropivacaïne (20cc)

SUMMARY:
Total knee replacement is a painful procedure. Many solutions have been proposed to diminish the post-operative doses of narcotics, including nerve blocks.

The purpose of the study is to compare if the adjunction of intra-articular ropivacaine to a femoral block is more effective on narcotics consumption than the block alone after TKR.

ELIGIBILITY:
Inclusion Criteria:

* Primary total knee replacement
* Age > 18 years old
* Accept the study

Exclusion Criteria:

* Revision surgery
* Use of anticoagulants drugs
* Neurologic disorder
* Unable to sign consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Narcotic consumption per 24 hours after surgery (mg/kg) | 48 hours

SECONDARY OUTCOMES:
VAS score at 24 hours | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dr Stéphane Pelet, MD,PhD, Principal Investigator — Hôpital Enfant-Jésus
Locations (1):
- CHA-Pavillon Enfant-Jésus, Québec, Quebec, Canada